CLINICAL TRIAL: NCT03793049
Title: Repeatability and Reproducibility of the CADence™System
Acronym: SEQUEL
Status: Completed | Type: Observational
Sponsor: AUM Cardiovascular, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 1030-002-03
Record Dates: First submitted 2019-01-02; First posted 2019-01-04 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-01

CONDITIONS: Coronary Artery Disease
Keywords: acoustic; ECG
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: CADence testing will be performed — CADence is a noninvasive, handheld device comprised of acoustic and ECG technology and software

SUMMARY:
This study is designed as a prospective study to capture data for evaluating the repeatability and reproducibility of the CADence™ System. The study will be conducted at 3 different study sites using 6 CADence™ systems. Each subject will be tested 4 separate times by 2 different operators at each site and will be tested at all 3 site locations in order to accomplish this evaluation. The study will enroll a total of at least 24 CADence positive patients and at least 24 CADence negative patients.

DETAILED DESCRIPTION:
The CADence™ system is comprised of a digital stethoscope used to record cardiac (heart) sounds, with integrated sensor used to record electrical activity of the heart (ECG), a single-use patient booklet, and the CADence™ Software application. CADence™ Software is a clinical decision support tool for the noninvasive functional evaluation of patients presenting with chest pain and at least two coronary artery disease risk factors that is intended to aid a qualified clinician's analysis of normal/physiological and pathological heart murmurs and in ruling out significant coronary disease as a cause for these symptoms of cardiovascular disease, utilizing simultaneous recording of cardiac sounds and ECG.

The purpose of this study is to assess the precision of the CADence site using multiple operators, cadence systems and clinical sites.

ELIGIBILITY:
Inclusion Criteria:

Subjects clinically indicated for nuclear stress test and who satisfy all the inclusion and exclusion criteria are eligible for participation.

Inclusion criteria:

1. Age 22 years or older
2. Willing and able to give informed consent
3. Clinical indication for nuclear stress test evaluation
4. Chest pain syndrome
5. Two or more coronary artery disease risk factors as defined by:

   * Dyslipidemia: LDL >130 mm/dL or HDL <35 mm/dL or on treatment for dyslipidemia
   * Hypertension: blood pressure >140 mmHg systolic, >90 mmHg diastolic or on blood pressure altering treatment
   * Obesity: BMI>28
   * Current cigarette smoking
   * Diabetes: Type 1 or 2
   * Family history: coronary disease in a first or second degree relative

Exclusion Criteria:

* Subjects clinically indicated for nuclear stress test and who satisfy all the inclusion and exclusion criteria are eligible for participation.

Inclusion criteria:

1. Age 22 years or older
2. Willing and able to give informed consent
3. Clinical indication for nuclear stress test evaluation
4. Chest pain syndrome
5. Two or more coronary artery disease risk factors as defined by:

   * Dyslipidemia: LDL >130 mm/dL or HDL <35 mm/dL or on treatment for dyslipidemia
   * Hypertension: blood pressure >140 mmHg systolic, >90 mmHg diastolic or on blood pressure altering treatment
   * Obesity: BMI>28
   * Current cigarette smoking
   * Diabetes: Type 1 or 2
   * Family history: coronary disease in a first or second degree relative

Exclusion criteria:

1. Body Mass Index (BMI)<18.5 or BMI >40
2. Known coronary disease as defined as:

   * Prior bypass surgery or coronary stenting
   * Q-wave infarction on a past EKG (>0.01 sec Q-wave duration in two adjacent leads)
3. Presence of pacemaker/defibrillator
4. Presence of artificial valve
5. Presence of obvious cyanotic or pre-diagnosed congenital heart defect and coarctation of the aorta
6. The presence of murmurs including moderate to severe valve disease, ventricular septal defects, and AV fistulae
7. Presence of moderate or severe valve disease as defined by >1/6 heart murmur on physical diagnosis
8. Left Ventricular Assist Device (LVAD)
9. Presence of scars on the site thorax areas
10. Participation in trial within 30 days prior to collecting CADenceTM data except participation in registry studies
11. Asthma with wheezing
12. Inability to lie flat in the supine position
13. Acute coronary syndrome with elevated cardiac biomarkers (TP>3x upper limit of normal (ULN) or CKMB>3x ULN)
14. Heart transplant
15. Current cocaine use (within the past 24 hours, as reported by subject)
16. Chronic Obstructive Pulmonary Disease (COPD)
17. Patient is not an acceptable candidate for CT angiography:

    * Renal failure with GFR <50
    * Iodinated contrast allergy
    * Elevated heart rate which cannot be controlled sufficiently to achieve a good CT angiogram
    * Body weight >350lbs
    * Persistent sinus rhythm abnormalities (e.g., atrial fibrillation) based on medical history.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with chest pain and 2 or more coronary artery disease risk factors
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-06-26 (Actual)

PRIMARY OUTCOMES:
Positive Percent Agreement and Negative Percent Agreement | 14 days
  repeatability and reproducibility

CONTACTS AND LOCATIONS:
Overall Officials: ROBERT WILSON, MD, Principal Investigator — University of Minnesota
Locations (3):
- United States (3):
  - 910 Medical, Minneapolis, Minnesota
  - Northfield Urgent Care Clinic, Northfield, Minnesota
  - Pivot Point Medical, Northfield, Minnesota

IPD SHARING:
Plan to Share IPD: No
WILL NOT BE SHARED

REFERENCES:
- [Background] Neglia D, Rovai D, Caselli C, Pietila M, Teresinska A, Aguade-Bruix S, Pizzi MN, Todiere G, Gimelli A, Schroeder S, Drosch T, Poddighe R, Casolo G, Anagnostopoulos C, Pugliese F, Rouzet F, Le Guludec D, Cappelli F, Valente S, Gensini GF, Zawaideh C, Capitanio S, Sambuceti G, Marsico F, Perrone Filardi P, Fernandez-Golfin C, Rincon LM, Graner FP, de Graaf MA, Fiechter M, Stehli J, Gaemperli O, Reyes E, Nkomo S, Maki M, Lorenzoni V, Turchetti G, Carpeggiani C, Marinelli M, Puzzuoli S, Mangione M, Marcheschi P, Mariani F, Giannessi D, Nekolla S, Lombardi M, Sicari R, Scholte AJ, Zamorano JL, Kaufmann PA, Underwood SR, Knuuti J; EVINCI Study Investigators. Detection of significant coronary artery disease by noninvasive anatomical and functional imaging. Circ Cardiovasc Imaging. 2015 Mar;8(3):e002179. doi: 10.1161/CIRCIMAGING.114.002179. PMID 25711274